CLINICAL TRIAL: NCT02015624
Title: EmploYEd Antithrombotic Therapies in Patients With Acute Coronary Syndromes HOspitalized in iTalian CCUs Registry
Brief Title: EYESHOT (EmploYEd Antithrombotic Therapies in Patients With Acute Coronary Syndromes HOspitalized in iTalian Coronary Care Units)
Acronym: EYESHOT
Status: Completed | Type: Observational
Sponsor: Heart Care Foundation (Other)
Collaborators: Centro Servizi ANMCO S.r.l. (Unknown); AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: EYESHOT
Record Dates: First submitted 2013-12-09; First posted 2013-12-19 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2014-03

CONDITIONS: Acute Coronary Syndromes
Keywords: Acute coronary syndromes; Intensive Care Unit
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This register will evaluate the use of different antithrombotic therapies, combinations of different drugs routinely used during any stage of hospital admission, with their timing, dosage and mode of administration, in patients with a diagnosis of Acute Coronary Syndrome in the Italian Coronary Care Unit during a study period of three weeks

ELIGIBILITY:
Inclusion criteria:

* All consecutive patients discharged with a diagnosis of Acute Coronary Syndrome ( Non ST elevation or ST Elevation) undergoing myocardial revascularization or conservative treatment , admitted to the Coronary Care Unit during the observation period established.
* Age ≥ 18 years
* Signed informed consent

Exclusion criteria:

* Patients enrolled in clinical trials of intervention
* Diagnosis of Acute Coronary Syndrome caused by confounding comorbidities (eg . Trauma or surgery after non- cardiac )
* Patients already enrolled in eyeshot from another center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of Acute Coronary Syndrome consecutively admitted in the Italian Cardiac Care Unit, located in hospitals with and without cardiac cath lab and cardiac surgery, during a period of 3 weeks
Sampling Method: Probability Sample
Enrollment: 2597 (Actual)
Dates: Start 2013-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Antithrombotic drugs in patient undergoing percutaneous transluminal coronary angiography, coronary artery bypass graft or no coronary revascularization | Participants will be followed for the duration of hospital stay, an expected average period of 7 days

SECONDARY OUTCOMES:
In-hospital ischemic and hemorrhagic events | Participants will be followed for the duration of hospital stay, an expected average period of 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Stefano De Servi, MD, Study Chair — Ospedale Civile - Legnano; Leonardo De Luca, MD, Study Chair — European Hospital - Roma
Locations (203):
- Italy (203):
  - Ospedale San Giovanni Di Dio, S.C. Cardiologia, Agrigento, AG
  - Ospedale Barone Lombardo, Cardiologia E Utic, Canicattì, AG
  - Ospedali Riuniti, Sod Cardiologia Ospedaliera E Utic, Ancona, AN
  - Istituto Scientifico Inrca, Uo Cardiologia/Utic/Telecardiologia, Ancona, AN
  - Ospedali Riuniti, U.O. Di Cardiologia, Iesi, AN
  - Ospedale Generale Regionale - Po U. Parini - U.O. Cardiologia E Cure Intensive Card., Aosta, AO
  - Ospedale Civile Ss. Filippo E Nicola, U.O. Cardiologia E Utic, Avezzano, AQ
  - Ospedale San Donato, U.O. Cardiologia, Arezzo, AR
  - Ospedale Miulli, U.O.C. Cardiologia - Utic, Acquaviva delle Fonti, BA
  - Ospedale San Paolo, Cardiologia-Utic, Bari, BA
  - Ospedale Consorziale Policlinico, U.O. Cardiologia Universitaria, Bari, BA
  - Ospedale Consorziale Policlinico, U.O. Di Cardiologia Ospedaliera, Bari, BA
  - Ospedale Di Venere, U.O.C. Di Cardiologia, Carbonara di Bari, BA
  - Azienda Ospedaliera Papa Giovanni Xxiii, U.S.C. Di Cardiologia, Bergamo, BG
  - Iob - Policlinico San Pietro, U.O.C. Cardiologia E Utic, Ponte San Pietro, BG
  - Ospedale Degli Infermi, Divisione Di Cardiologia, Biella, BI
  - Ospedale Santa Maria Del Prato, U.O. Di Cardiologia, Feltre, BL
  - Ospedale Di Bentivoglio, U.O. Di Cardiologia, Bentivoglio, BO
  - Ospedale Maggiore, U.O. Di Cardiologia, Bologna, BO
  - Ospedale Nuovo S. Maria Della Scaletta, Uoc Cardiologia, Imola, BO
  - Ospedale Perrino, U.O.C. Di Cardiologia, Brindisi, BR
  - Spedali Civili, Cardiologia, Brescia, BS
  - Istituto Osped. Fondazione Poliambulanza, Unita' Operativa Di Cardiologia, Brescia, BS
  - Ospedale Civile Mellini - Divisione di Cardiologia, Chiari, BS
  - Ospedale Civile Di Valle Camonica, Divisione Di Cardiologia, Esine, BS
  - Ospedale Generale Regionale, Bolzano, BZ
  - Presidio Ospedaliero Ss Trinita', Sc Di Cardiologia, Cagliari, CA
  - Ospedale San Giovanni Di Dio, Cattedra E Divisione Di Cardiologia, Cagliari, CA
  - Azienda Ospedaliera G. Brotzu, Cagliari, CA
  - Ospedale A. Cardarelli, U.O. Cardiologia E Utic, Campobasso, CB
  - Ospedale San Timoteo, Uoc Clinica-Intensiva-Vascolare, Termoli, CB
  - Clinica Pineta Grande, Unita Terapia Intensiva Coronarica, Castel Volturno, CE
  - Ospedale San Giuseppe E Melorio, U.O.C. Cardiologia Utic, Santa Maria Capua Vetere, CE
  - Presidio Ospedaliero San Rocco, Emergenze Cardiologiche, Sessa Aurunca, CE
  - Ospedale Policlinico Ss. Annunziata, Cardiologia-Utic, Chieti, CH
  - Ospedale San Pio Da Pietrelcina, Cardiologia, Vasto, CH
  - Az. Ospedaliera Vittorio Emanuele Iii, S.C. Cardiologia - Utic, Gela, CL
  - Ospedale Regina Montis Regalis, U.O. Cardiologia-Utic, Mondovì, CN
  - Ospedale Maggiore Ss. Annunziata, Sc Cardiologia, Savigliano, CN
  - Ospedale Generale Di Zona Valduce, Unita' Operativa Di Cardiologia, Como, CO
  - Ospedale Sacra Famiglia Fbf, Unita' Operativa Di Cardiologia, Erba, CO
  - Ospedale Moriggia Pelascini, Unita' Operativa Di Cardiologia, Gravedona, CO
  - Ospedale S. Anna, U.O.C. Di Cardiologia, San Fermo della Battaglia, CO
  - Ospedale Civile Oglio Po, U.O. Di Cardiologia-Utic, Casalmaggiore, CR
  - Istituti Ospitalieri - UO Cardiologia, Cremona, CR
  - Ospedale Civile Ferrari, U.O.C. Cardiologia-Utic-Emodinamica, Castrovillari, CS
  - Ospedale Santissima Annunziata, Uoc Cardiologia, Cosenza, CS
  - Spoke Cetraro-Paola, U.O. Cardiologia E Utic, Paola, CS
  - Ospedale Civile N. Giannettasio, U.O. Cardiologia E Utic, Rossano, CS
  - P. O. Gravina E Santo Pietro, U.O. Di Cardiologia-Utic, Caltagirone, CT
  - P.O. Garibaldi Centro, U.O.C. Cardiologia, Catania, CT
  - P.O. Ospedale Ferrarotto-Alessi, U.O. Clinicizzata Di Cardiologia, Catania, CT
  - Az Ospedaliera Universitaria Materdomini, U.O. Cardiologia - Campus Universitario, Catanzaro, CZ
  - Ospedale Civile Pugliese, Utic-Emodinamica E Card. Interventistica, Catanzaro, CZ
  - Ospedale M.Bufalini, U.O. Di Cardiologia-Utic, Cesena, FC
  - Ospedale G.B. Morgagni - L. Pierantoni, U.O. Cardiologia, Forlì, FC
  - Ospedale Ss. Annunziata, U.O. Di Cardiologia, Cento, FE
  - Ospedale Del Delta, U.O. Cardiologia, Lagosanto, FE
  - Ospedale Civile Giuseppe Tatarella, U.O. Di Cardiologia - Utic, Cerignola, FG
  - Ospedali Riuniti, S.C. Di Cardiologia Univ.-Utic, Foggia, FG
  - Ospedale casa Sollievo della Sofferenza - Cardiologia - UTIC, San Giovanni Rotondo, FG
  - Ospedale Padre Antero Micone, Cardiologia - Utic, Genova, GE
  - Irccs San Martino Ist Ricerca Sul Cancro, Unita' Operativa Cardiologia, Genova, GE
  - Ospedale Civile San Polo, S.O.C. Cardiologia, Monfalcone, GO
  - Ospedale della Misericordia - UO Cardiologia, Grosseto, GR
  - Presidio Ospedaliero, U.O. Cardiologia, Sanremo, IM
  - Ospedale Civile San Giovanni Di Dio, U.O. Cardiologia, Crotone, KR
  - Ospedale Alessandro Manzoni - SC di Cardiologia, Lecco, LC
  - Ospedale San Leopoldo Mandic, Cardiologia - Ucc, Merate, LC
  - Presidio Ospedaliero F. Ferrari, Cardiologia - Utic, Casarano, LE
  - Ospedale San Giuseppe Da Copertino, U.O. Di Cardiologia-Utic, Copertino, LE
  - Ospedale Civile Sacro Cuore Di Gesu', Uo Cardiologia Utic, Gallipoli, LE
  - Citta' Di Lecce Hospital, U.O. Di Cardiologia, Lecce, LE
  - Ospedale Vito Fazzi, U.O. Di Cardiologia, Lecce, LE
  - Ospedale Cardinale Panico - U.O. Cardiologia UTIC, Tricase, LE
  - Ospedale Villamarina, Cardiologia E Utic, Piombino, LI
  - Ospedale Civico, Cardiologia 2, Codogno, LO
  - Ospedale Santa Croce, Ss Di Cardiologia, Castelnuovo di Garfagnana, LU
  - Nuovo Ospedale Versilia, Sc Cardiologia, Lido di Camaiore, LU
  - Ospedale Campo Di Marte, U.O. Di Cardiologia, Lucca, LU
  - Ospedale San Gerardo, U.O. Cardiologia-Utic, Monza, MB
  - Policlinico Di Monza, Uo Cardiol. Clinica E Scompenso Cardiaco, Monza, MB
  - P.O. Sant'Agata Di Militello, U.O. Cardiologia -Utic, Sant'Agata di Militello, ME
  - Ospedale Di Cernusco Sul Naviglio, U. O. Di Cardiologia E Ucc, Cernusco sul Naviglio, MI
  - Ospedale Bassini, U.O. Cardiologia E Utic, Cinisello Balsamo, MI
  - Ospedale Civile, Utic - Cardiologia, Legnano, MI
  - Ospedale Civile Fornaroli, U.O. Cardiologia, Magenta, MI
  - Ospedale Fatebenefratelli e Oftalmico - Cardiologia e UCC, Milan, MI
  - Ospedale Maggiore Policlinico, Divisione Di Cardiologia, Milan, MI
  - Istituto Clinico Citta' Studi, U.O. Cardiologia, Milan, MI
  - Centro Cardiologico Monzino - Terapia Intensiva Cardiologica UTIC, Milan, MI
  - Ospedale San Paolo, Divisione Di Cardiologia, Milan, MI
  - Ospedale San Luca-Centro Auxologico, U.O. Cardiologia, Milan, MI
  - Ospedale L. Sacco, Divisione Di Cardiologia, Milan, MI
  - Ospedale Niguarda, Cardiologia 1 - Emodinamica, Milan, MI
  - Irccs Policlinico Multimedica, U.O. Cardiologia/Ucc, Sesto San Giovanni, MI
  - Ospedale Di Vizzolo Predabissi, Uo Cardiologia E Ucc, Vizzolo Predabissi, MI
  - Ospedali Destra Secchia, Cardiologia E Utic, Pieve di Coriano, MN
  - Ospedale Madonna Delle Grazie, U.O. Cardiologia-Utic-Angiologia, Matera, Mount
  - Ospedale Giovanni Paolo Ii, Cardiologia Utic, Policoro, Mount
  - Nuovo Ospedale Sant'Agostino-Estense, U.O. Di Cardiologia, Modena, MO
  - Ftgm - Stabilimento Di Massa, U.O. Cardiologia Adulti, Massa, MS
  - Ospedale Ss. Giacomo E Cristoforo, U.O. Cardiologia-Utic, Massa, MS
  - Ospedale San Francesco, Cardiologia - Utic, Nuoro, NU
  - Ospedale Giovanni Paolo Ii, Utic - Cardiologia, Olbia, OT
  - Fondazione San Raffaele G. Giglio, U.O. Cardiologia E Utic, Cefalù, PA
  - Osp. Buccheri La Ferla Fatebenefratelli, Cardiologia - Utic, Palermo, PA
  - Arnas P.O. Civico E Benfratelli, U.O. Cardiologia, Palermo, PA
  - Aor Villa Sofia-Cervello P.O. Cervello, U.O. Cardiologia, Palermo, PA
  - Aor Villa Sofia-Cervello Po Villa Sofia, U.O.C. Cardiologia E Utic, Palermo, PA
  - Ospedale Civico, U.O. Cardiologia, Partinico, PA
  - Ospedale Di Camposampiero, U.O.A. Cardiologia, Camposampiero, PD
  - Ospedale Di Cittadella, U.O. Cardiologia, Cittadella, PD
  - Ospedale Di Este, U.O.C. Cardiovascolare, Este, PD
  - Azienda Ospedaliera Padova, Clinica Cardiologica, Padua, PD
  - Ospedale Civile Immacolata Concezione, Cardiologia E Utic, Piove di Sacco, PD
  - Ospedale Civile Dello Spirito Santo, Utic E Cardiologia Interventistica, Pescara, PE
  - Presidio Ospedaliero Citta' Di Castello, U.O. Di Cardiologia, Città di Castello, PG
  - Nuovo Ospedale San Giovanni Battista, S.C. Cardiologia, Foligno, PG
  - Azienda Ospedaliera di Perugia, Perugia, PG
  - Ftgm - Stabilimento Di Pisa, Cardiologia E Medicina Cariovascolare, Pisa, PI
  - Azienda Ospedaliera S.Maria Degli Angeli, S.O.C. Cardiologia, Pordenone, PN
  - Ospedale Civile, U.O.C. Cardiologia - Utic, Fidenza, PR
  - Azienda Ospedaliera San Salvatore, U.O.S.D. Unita' Coronarica, Pesaro, PU
  - Ospedale Santa Maria Della Misericordia, Cardiologia - Utic, Urbino, PU
  - Fondazione IRCCS Policlinico San Matteo - Card. con UCC-Lab. Ricerca Sperim. Card., Pavia, PV
  - Ospedale Civile, Cardiologia, Vigevano, PV
  - Ospedale Civile, U.O. Di Cardiologia, Lugo, RA
  - Ospedale Civile Santa Maria Delle Croci, U.O. Di Cardiologia, Ravenna, RA
  - Ospedale Civile, U.O. Cardiologia-Utic, Locri, RC
  - Ospedali Riuniti G. Melacrino F. Bianchi, Divisione Di Cardiologia, Reggio Calabria, RC
  - Ospedale Civile, U.O.C. Di Cardiologia, Guastalla, RE
  - Arcispedale Santa Maria Nuova - UO Degenza Cardiologica, Reggio Emilia, RE
  - Ospedale Riccardo Guzzardi, U.O.C. Di Cardiologia, Vittoria, RG
  - P.O. San Camillo de Lellis, U.O. Cardiologia Complessa Con Utic, Rieti, RI
  - Ospedali Riuniti Albano-Genzano, U.O.C. Di Cardiologia E Utic, Albano Laziale, RM
  - Ospedali Riuniti Anzio-Nettuno, U.O. Di Cardiologia, Anzio, RM
  - Ospedale L. Parodi Delfino, U.O. Complessa Di Cardiologia, Colleferro, RM
  - Ospedale San Filippo Neri, Uoc Cardiologia E Utic, Roma, RM
  - Ospedale San Camillo, Uoc Cardiologia I, Roma, RM
  - Ospedale Sandro Pertini, Uosd Terapia Intensiva Cardiologica, Roma, RM
  - Casa Di Cura Nuova Itor, Reparto Di Cardiologia E Utic, Roma, RM
  - Policlinico Umberto Primo, Cardiologia B - Cardiologia E Angiologia, Roma, RM
  - Aurelia Hospital, U.O.C Cardiologia, Roma, RM
  - Policlinico Casilino, U.O. Cardiologia, Roma, RM
  - Ospedale Madre Giuseppina Vannini, U.O.C. Cardiologia, Roma, RM
  - Ao San Giovanni Addolorata, Ao San Giovanni Addolorata Cardiologia Ii, Roma, RM
  - Ospedale Fatebenefratelli, U.O.C. Cardiologia, Roma, RM
  - Ospedale San Pietro Fatebenefratelli, U.O Complessa Di Cardiologia, Roma, RM
  - Ospedale Sant'Andrea Di Roma, U.O.C. Cardiologia, Roma, RM
  - Ospedale Infermi - UO Cardiologia, Rimini, RN
  - Ospedale S. Maria Regina Degli Angeli, U.O. Cardiologia, Adria, RO
  - Ospedale Santa Maria Della Misericordia, U.O.C. Cardiologia, Rovigo, RO
  - Presidio Osped. S. Maria Della Speranza, U.O. Di Cardiologia, Battipaglia, SA
  - Ospedale Maria Ss. Addolorata, U.O. Di Cardiologia, Eboli, SA
  - A.O.U.S. Giovanni Di Dio-Ruggi D'Aragona, U.O.C. Utic, Salerno, SA
  - Ospedale Valdichiana, Cardiologia E Utic, Montepulciano, SI
  - Ospedale G. Di Maria, Cardiologia Utic, Avola, SR
  - P.O. Lentini, U.O. Di Cardiologia Con Utic, Lentini, SR
  - Azienda Ospedaliera Umberto I, U.O. Di Cardiologia, Syracuse, SR
  - Ospedale Civile M. Giannuzzi, Cardiologia E Utic, Manduria, TA
  - Ospedale S. Giuseppe Moscati, S.C. Cardiologia, Taranto, TA
  - Ospedale Ss. Annunziata, S.C. Cardiologia-Utic, Taranto, TA
  - Ospedale Civile G. Mazzini, U.O. Cardiologia - Utic, Teramo, TE
  - Ospedale Santa Maria Del Carmine, Divisione Di Cardiologia, Rovereto, TN
  - Ospedale Santa Chiara, Divisione Di Cardiologia, Trento, TN
  - Ospedale Molinette, S.C. Di Cardiologia 2, Torino, TO
  - Ospedale Molinette, S.C.D.U. Cardiologia 1, Torino, TO
  - Ospedale Martini - U.O. Cardiologia/UTIC, Torino, TO
  - Ospedale Giovanni Bosco, Sc Cardiologia, Torino, TO
  - Osp. Ajello C/O Osp. Vittorio Emanueleii, U.O. Cardiologia, Castelvetrano, TP
  - Ospedale Civile Sant'Antonio Abate, U.O.C. Di Cardiologia E Utic, Erice, TP
  - Presidio Ospedaliero Paolo Borsellino, U.O. Cardiologia- Utic, Marsala, TP
  - Azienda Ospedaliera Santa Maria, S.C. Di Cardiologia, Terni, TR
  - Aou Ospedali Riuniti, S.O.C. Cardiologia - Ospedale Cattinara, Trieste, TS
  - Ospedale Ca' Foncello, U.O.C. Cardiologia, Treviso, TV
  - Aou Santa Maria Della Misericordia, S.O.C. Cardiologia, Udine, UD
  - Ospedale Di Circolo Di Busto Arsizio, Divisione Di Cardiologia, Busto Arsizio, VA
  - Ospedale S. Antonio Abate, U.O. Di Cardiologia, Gallarate, VA
  - Presidio Ospedaliero Di Saronno, U.O.C. Di Cardiologia, Saronno, VA
  - Ospedale Di Circolo Galmarini, Cardiologia, Tradate, VA
  - Ospedale Di Circolo E Fondazione Macchi, Ssd Unita' Di Cure Intensive Coronariche, Varese, VA
  - Ospedale Civile, U.O.C. Cardiologia, Chioggia, VE
  - Ospedale Dell'Angelo, U.O. Cardiologia, Mestre, VE
  - Ospedale Civile Di Venezia, U.O. Di Cardiologia, Venezia, VE
  - Ospedale San Bassiano, Struttura Complessa Di Cardiologia, Bassano del Grappa, VI
  - Ospedale Unico Ulss 4, U.O.C. Cardiologia - Ucic, Santorso, VI
  - Ospedale Mater Salutis, U.O.C. Cardiologia, Legnago, VR
  - Casa Di Cura Dr. Pederzoli, Servizio Di Cardiologia, Peschiera del Garda, VR
  - Ospedale G. Fracastoro, U.O.C. Di Cardiologia, San Bonifacio, VR
  - Azienda Ospedaliera G. Rummo, Benevento
  - Ospedale Ss. Trinita', S.C. Di Cardiologia, Borgomanero
  - Ospedale Generale Di Zona, U.O. Cardiologia - Utic, Giugliano in Campania
  - Clinica Mediterranea, U.O. Di Cardiologia, Napoli
  - AORN Cardarelli - UO SC Cardiologia con UTIC, Napoli
  - Aorn Osp. Dei Colli- Po Vincenzo Monaldi, U.O.C. Cardiologia - S.U.N., Napoli
  - Aorn Osp. Dei Colli- Po Vincenzo Monaldi, U.O.C. Cardiologia, Napoli
  - Aou Federico Ii, Utic, Napoli
  - Ospedale Dei Pellegrini, Uoc Cardiologia-Utic, Napoli
  - Ospedale Loreto Mare, U.O. Cardiologia Con Utic, Napoli
  - Pres. Ospedaliero S. Maria Della Pieta', U.O. Cardiologia E Utic, Nola
  - AO Univ. Maggiore della Carità - Cardiologia 2, Novara
  - Ospedale Santa Maria Delle Grazie, U.O. Cardiologia - Utic, Pozzuoli

REFERENCES:
- [Background] De Luca L, Leonardi S, Smecca IM, Formigli D, Lucci D, Gonzini L, Tuccillo B, Olivari Z, Gulizia MM, Bovenzi FM, De Servi S; EYESHOT Investigators. Contemporary antithrombotic strategies in patients with acute coronary syndromes managed without revascularization: insights from the EYESHOT study. Eur Heart J Cardiovasc Pharmacother. 2015 Jul;1(3):168-78. doi: 10.1093/ehjcvp/pvv006. Epub 2015 Feb 24. PMID 27533991
- [Background] De Luca L, Musumeci G, Leonardi S, Gonzini L, Cavallini C, Calabro P, Mauro C, Cacciavillani L, Savonitto S, De Servi S; EYESHOT Investigators. Antithrombotic strategies in the catheterization laboratory for patients with acute coronary syndromes undergoing percutaneous coronary interventions: insights from the EmploYEd antithrombotic therapies in patients with acute coronary Syndromes HOspitalized in iTalian cardiac care units Registry. J Cardiovasc Med (Hagerstown). 2017 Aug;18(8):580-589. doi: 10.2459/JCM.0000000000000533. PMID 28639987
- [Background] De Luca L, Pennacchi M, Musumeci G, D'Ascenzo F, Gallo P, Rigattieri S, Granatelli A, Berti S, Gulizia MM, De Servi S, Bolognese L; a nome dei Ricercatori EYESHOT e SCOPE. [Temporal evolution of antithrombotic therapy use in patients with acute coronary syndromes undergoing percutaneous coronary intervention in Italy: comparison between the EYESHOT and SCOPE registries]. G Ital Cardiol (Rome). 2018 Feb;19(2):101-110. doi: 10.1714/2868.28941. Italian. PMID 29531382
- [Result] De Luca L, Leonardi S, Cavallini C, Lucci D, Musumeci G, Caporale R, Abrignani MG, Lupi A, Rakar S, Gulizia MM, Bovenzi FM, De Servi S; EYESHOT Investigators. Contemporary antithrombotic strategies in patients with acute coronary syndrome admitted to cardiac care units in Italy: The EYESHOT Study. Eur Heart J Acute Cardiovasc Care. 2015 Oct;4(5):441-52. doi: 10.1177/2048872614560505. Epub 2014 Nov 20. PMID 25414322
- [Derived] De Luca L, Leonardi S, Tubaro M, Gonzini L, Lucci D, Trimarco B, Misuraca G, Ledda A, Gulizia MM, De Servi S; EYESHOT Investigators. Is the use of risk scores an indicator of guideline adherence for patients with acute coronary syndromes? Insights from the EYESHOT Registry. Int J Cardiol. 2015;187:80-3. doi: 10.1016/j.ijcard.2015.03.343. Epub 2015 Mar 24. No abstract available. PMID 25828318